CLINICAL TRIAL: NCT06892288
Title: A Phase 2b, Multicenter, Double-blind, Randomized, Placebo Controlled Study to Assess the Efficacy and Safety of Weekly Doses of GLM101 Administered Intravenously to Participants With PMM2-CDG (POLAR Trial)
Brief Title: A Study to Assess the Efficacy and Safety of Weekly Doses of GLM101 in Participants With PMM2-CDG
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Glycomine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLM101-003
Record Dates: First submitted 2025-02-06; First posted 2025-03-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Phosphomannomutase 2 Deficiency; PMM2-CDG
Keywords: GLM101; CDG; CDG 1a; PMM2; Ataxia; GLM101-003
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A; Ataxia | interventions — Double-Blind Method

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either GLM101 or placebo (Part A) and subsequently all participants will receive GLM101 (Part B).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLM101- 30 mg/kg weekly administered IV in Part A (double-blind) and Part B (open-label) (Experimental)
  Interventions: Drug: GLM101 (Part A, Double-blind); Drug: GLM101 (Part B, Open-label)
- Placebo weekly admin. IV in Part A (double-blind); 30 mg/kg weekly admin. IV in Part B (open-label) (Placebo Comparator)
  Interventions: Drug: Placebo (Part A, Double-blind); Drug: GLM101 (Part B, Open-label)

INTERVENTIONS:
Drug: GLM101 (Part A, Double-blind) — IV infusions, 30 mg/kg once weekly for 24 weeks, for participants randomized to GLM101 in Part A
  Arms: GLM101- 30 mg/kg weekly administered IV in Part A (double-blind) and Part B (open-label)
Drug: Placebo (Part A, Double-blind) — IV infusions, 30 mg/kg once weekly for 24 weeks, for participants randomized to Placebo in Part A
  Arms: Placebo weekly admin. IV in Part A (double-blind); 30 mg/kg weekly admin. IV in Part B (open-label)
Drug: GLM101 (Part B, Open-label) — IV infusions, 30 mg/kg once weekly from week 25 to 48, to all participants

SUMMARY:
This study is evaluating the safety, effectiveness, and how the body absorbs, distributes, and eliminates GLM101, for participants with PMM2-CDG, including children, adolescents, and adults. Researchers will compare participants receiving GLM101 to those receiving a placebo to see if GLM101 improves symptoms of PMM2-CDG.

The study includes two treatment parts: a 24-week double blind placebo-controlled treatment period (Part A), and a 24-week open-label phase where every participant will receive GLM101(Part B).

DETAILED DESCRIPTION:
This Phase 2b, multicenter, randomized, double-blind, placebo-controlled clinical study is designed to evaluate the efficacy, safety, and pharmacokinetics (PK) of GLM101 in adult, adolescent, and pediatric participants with PMM2-CDG. The study is structured into: a 4-week Screening Period, a 24-week Double-blind Treatment Period (Part A) to assess primary efficacy, a 24-week Open-label Extension Period (Part B), and a safety follow-up visit conducted 4 weeks after the last infusion. In Part A, participants will be randomly assigned to receive weekly intravenous infusions of either GLM101 at 30 mg/kg or a placebo for 24 weeks. After the end of Part A, participants will transition into Part B, a 24-week open-label extension where all participants will receive GLM101. The primary objective of the trial is to identify changes from baseline in coordination and muscle movement (ataxia) using the International Co-operative Ataxia Rating Scale (ICARS) after 24 weeks of taking GLM101 compared to a placebo in PMM2-CDG patients.

ELIGIBILITY:
Inclusion criteria: Participant is eligible for participation in the study if all of the following apply:

* Participant is aged ≥ 4 years old at the time of signing the consent.
* Participant with molecular diagnosis of PMM2-CDG. Diagnosis is defined as biallelic pathogenic and/or likely pathogenic variants, or, in the case of variants of uncertain pathogenicity, demonstration of biallelic variants and PMM2 enzyme activity consistent with a diagnosis of PMM2-CDG. Diagnosis with laboratory report(s) on file is required.
* Participant is willing and capable of completing the ICARS in its entirety without any assessment deemed as "not evaluable".
* Participant screening total ICARS score is ≥ 20 and ≤ 80 .
* Male or female participant has appropriate measures in place to prevent pregnancy:

  * If the participant is a woman of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile (permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy), she must not be pregnant (confirmed by a negative serum pregnancy test), is using a medically accepted method of contraception (abstinence, a hormonal contraceptive associated with inhibition of ovulation in conjunction with a barrier method, or use of an intrauterine device), and must agree to continue using this method for 50 days after the last infusion. Note: sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception.
  * If the participant is a female of non-childbearing potential, she must be premenarchal, surgically sterile, or must have an ovarian dysfunction confirmed by a follicle stimulating hormone > 40 IU/ L (or higher per local institutional guidelines) and absence of menses for 12 months after last menstrual bleeding without an alternative medical cause.
  * If the participant is a sexually active male with female partners, the participant agrees to use a medically acceptable method of contraception (abstinence, the partner taking a hormonal contraceptive in conjunction with male participant using male condom, or use by the partner of an intrauterine device with a male participant using male condom) and agrees to continue using this method for 50 days after the last infusion.
* If the participant is male, he must agree to refrain from donating sperm during the study and 50 days after the last infusion.
* The participant is willing and able to provide informed consent/assent, directly or through his/her legally authorized representative.
* The participant has a caregiver who is willing and able to complete questionnaires and provide informed consent.

Exclusion criteria: Participant will be excluded from participation in the study if any of the following criteria apply:

* Has uncontrolled cardiovascular, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric or other significant disease based on the investigator judgment.
* Diagnosis of congenital disorder of glycosylation (CDG) other than PMM2; Diagnosis is defined as biallelic pathogenic and/or likely pathogenic variants, or, in the case of variants of uncertain pathogenicity, demonstration of biallelic variants and the defined CDG enzyme activity consistent with a diagnosis of the CDG other than PMM2 CDG.
* Has a history of liver transplant.
* Has an active infection requiring parenteral antibiotics, antivirals, antifungals or treatment with systemic steroids within 7 days prior to screening.
* Has a history of drug or alcohol use disorder within 12 months prior to screening.
* Has had a major surgical procedure within 30 days prior to screening or an upcoming planned major surgery.
* Previous history of GLM101 administration.
* Is currently participating in another interventional clinical study or has completed another clinical study with an investigational drug or device within 30 days or 5 half-lives (whichever is longer) before enrollment.
* Have consumed products or supplements containing mannose or biotin within 2 weeks prior to screening.
* Elevated liver function tests: ALT or AST > 3 × ULN OR total bilirubin > 2 × ULN or international normalized ratio (INR) > 1.5 (if no anti-coagulation treatment) or INR > 4 (if participant on anti-coagulation treatment).
* Has screening laboratory value(s) considered clinically significant and not related to PMM2-CDG based on the investigator judgment.
* Has serology positive for hepatitis B surface antigen or hepatitis C antibody during screening.
* Has a QT interval by Fridericia (QTcF) ≥ 450 ms, or other electrocardiogram abnormalities judged as clinically significant by the investigator.
* Has history or presence, upon clinical evaluation, of any illness that might impact the safety of GLM101 infusion or evaluability of drug effect based on the investigator's and Sponsor's Medical Monitor's discretion.
* Participant weighs above 120 kg.
* Participant has a known or suspected hypersensitivity to GLM101 or any components of the formulation used.
* Any other reason for which, in the investigator's opinion, makes the participant unsuitable for study participation.
* If female, must not be breastfeeding.
* Estimated glomerular filtration rate (eGFR) <45 mL/min/ 1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation for participants ≥ 18 years or Schwartz equation for participants <18 years of age at screening.
* Persons who have been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Ataxia Changes Using the International Cooperative Ataxia Rating Scale (ICARS) in PMM2-CDG Patients at 24 weeks | At baseline and at week 24.
  To characterize the change from Baseline in ataxia at 24 weeks, comparing GLM101 to placebo in participants with PMM2-CDG as assessed by ICARS. The scale is scored out of 100 with 19 items and four subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment (Part A).

SECONDARY OUTCOMES:
Evaluation of Change from Baseline in Gross Motor Function at 24 Weeks Using the Neuromuscular Gross Motor Outcome (GRO) in PMM2-CDG Patients | At baseline and at week 24.
  To characterize the change from Baseline in gross motor function at 24 weeks, comparing GLM101 to placebo in participants with PMM2-CDG as assessed by GRO. The GRO is a gross neuromuscular motor outcome measure designed to assess whole body strength, motor development, and function for all levels of ability across the lifespan (Part A).
Evaluation of Change from Baseline in Ataxia at 24 Weeks Using the Scale for the Assess and Rating of Ataxia (SARA) in PMM2-CDG Patients | At baseline and at week 24.
  To characterize the change from Baseline in ataxia at 24 weeks, comparing GLM101 to placebo in participants with PMM2-CDG as assessed by SARA. It consists of eight items of patient performance including gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide. It is scored out of 40 points with higher scores indicating higher levels of impairment (Part A).
Evaluation of Change in Global Impression of Improvement/Changes and Severity at 24 Weeks by PMM2-CDG Patients, Caregiver and Physician | At baseline and at week 24.
  To evaluate the participant, caregiver, and physician global impression of improvement/change and severity at 24 weeks, comparing GLM101 to placebo (Part A).
Reporting of Adverse Events (AEs) in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
Reporting of Blood Pressure in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
  Blood pressure will be measured in millimeters of mercury (mmHg).
Reporting of Body Temperature in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
  Body Temperature will be measured in degree Celsius (°C).
Reporting of Pulse Rate in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
  Pulse rate will be measured in beats per minute (bpm).
Reporting of Respiratory Rate in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
  Respiratory rate will be measured in breaths per minute.
Reporting of Cardiovascular Health Using Electrocardiogram (ECG) in PMM2-CDG Patients at 24 weeks (Part A) | At baseline and up to week 24.
  The following parameters will be evaluated: heart rate, PR, RR, QRS, QT intervals along with information on T and U-wave morphology.
Evaluation of Ataxia Changes Using the International Cooperative Ataxia Rating Scale (ICARS) in PMM2-CDG Patients from baseline to the End of the Study | At baseline and at weeks 24 and 48.
  To evaluate the effect of GLM101 on changes in ICARS score to the end of study. The objective is to evaluate ICARS changes over 48 weeks, comparing early versus delayed GLM101 treatment, placebo-to-GLM101 transitions, and visit-wise changes in participants receiving GLM101 (Part B).
Evaluation of Changes in the Neuromuscular Gross Motor Outcome (GRO) Score in PMM2-CDG Patients from baseline to the End of the Study | At baseline and at weeks 24 and 48.
  To evaluate the effect of GLM101 on changes in GRO score to the end of study. The objective is to evaluate changes in GRO score over 48 weeks, comparing early versus delayed GLM101 treatment, placebo-to-GLM101 transitions, and visit-wise changes in participants receiving GLM101 (Part B).
Evaluation of Changes in the Scale for the Assess and Rating of Ataxia (SARA) Score in PMM2-CDG Patients from baseline to the End of the Study | At baseline and at weeks 24 and 48.
  To evaluate the effect of GLM101 on change in SARA score to the end of study. The objective is to evaluate changes in SARA Score over 48 weeks, comparing early versus delayed GLM101 treatment, placebo-to-GLM101 transitions, and visit-wise changes in participants receiving GLM101 (Part B).
Evaluation of Change in Global Impression of Improvement/Changes and Severity from baseline to the End of the Study by PMM2-CDG Patients, Caregiver and Physician | At baseline and up to week 48.
  To evaluate the participant, caregiver, and physician global impression of improvement/change and severity up to 48 weeks of dosing with GLM101. Evaluation of visit-wise changes in participant, caregiver, and clinician impressions of change, severity, and improvement for overall, ataxia, and gross motor function (Part B).
Reporting of Adverse Events in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
Reporting of Blood Pressure in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
  Blood pressure will be measured in millimeters of mercury (mmHg).
Reporting of Pulse Rate in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
  Pulse rate will be measured in beats per minute (bpm).
Reporting of Body Temperature in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
  Body Temperature will be measured in degree Celsius (°C).
Reporting of Respiratory Rate in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
  Respiratory rate will be measured in breaths per minute.
Reporting of Cardiovascular Health Changes Using Electrocardiogram (ECG) in PMM2-CDG Patients from Baseline to the End of the Study (Part B) | At baseline and up to week 48.
  The following parameters will be evaluated: heart rate, PR, RR, QRS, QT intervals along with information on T and U-wave morphology.
Maximum Concentration (Cmax) of Mannose-1-phosphate (M1P) in PMM2-CDG Patients as Key PK Parameter over 48 weeks to the End of the Study (Part B) | At Baseline and at weeks 11, 12, 20, 21, 35, 36, 44, 45.
  Cmax will be estimated using Blood Samples collected Pre- and Post-Infusion.
Time from dosing to the Maximum Concentration (tmax) of Mannose-1-phosphate (M1P) in PMM2-CDG Patients as Key PK Parameter over 48 weeks to the End of the Study (Part B) | At Baseline and at weeks 11, 12, 20, 21, 35, 36, 44, 45.
  tmax will be estimated using Blood Samples collected Pre- and Post-Infusion.
Area under the concentration versus time curve (AUC) of Mannose-1-phosphate (M1P) in PMM2-CDG Patients as Key PK Parameter over 48 weeks to the End of the Study (Part B) | At Baseline and at weeks 11, 12, 20, 21, 35, 36, 44, 45.
  AUC will be estimated using Blood Samples collected Pre- and Post-Infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Glycomine, Inc.
Locations (15):
- United States (4):
  - University of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- UZ Leuven, Campus Gasthuisberg, Leuven, Belgium
- Vseobecna fakultni nemocnice v Praze, Prague, Czechia
- AP-HP Hopital Necker-Enfants Malades, Paris, France
- Universitaetsklinikum Muenster, Münster, Germany
- Italy (2):
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico-San Marco, Catania
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Instytut Matki i Dziecka, Warsaw, Poland
- Unidade Local de Saúde de Santo António, Porto, Portugal
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
- Birmingham Women's and Children's NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided